CLINICAL TRIAL: NCT03951961
Title: Midostaurin in MRD (Minimal Residual Disease) Positive Acute Myeloid Leukemia After Allogeneic Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient Recruitment
Sponsor: University of Jena (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Sebastian Scholl, PD Dr. med., Principal Investigator, University of Jena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAURITIUS; 2019-000136-26 (EudraCT Number)
Record Dates: First submitted 2019-05-09; First posted 2019-05-16 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Acute Myeloid Leukemia, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — midostaurin

STUDY DESIGN:
Intervention Model Description: single-arm, multicenter phase II, non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Midostaurin (Experimental): 50 mg Midostaurin bid for 12 months
  Interventions: Drug: Midostaurin

INTERVENTIONS:
Drug: Midostaurin — 50mg Midostaurin bid for 12 months

SUMMARY:
The MAURITIUS trial is a single-arm, multicenter phase II study of single treatment with midostaurin being applied to AML (acute myeloid leukemia) patients with activating FLT3 (FMS-like tyrosine kinase3) mutations and either molecular relapse or persistent molecular positivity after allogeneic SCT. The leukemia-free survival (LFS), the achievement of "MRD low" as well as the incidence of GvHD after transplantation reflect the most relevant endpoints of this non-randomized clinical trial.

DETAILED DESCRIPTION:
The clinical situation of AML (acute myeloid leukemia) relapse after intensive chemotherapy or even after allogeneic SCT represents a huge challenge in hematology. So far, no FLT3-TKI (Tyrosine kinase Inhibitor) has been approved for the treatment of relapsed or refractory AML with activating FLT3 mutations in the European Union.

For elderly and unfit patients at primary diagnosis and for patients with AML relapse after induction and consolidation chemotherapy (including those with allogeneic SCT) who are not eligible for any further intensive treatment approach, AML therapy with HMA (hypomethylating agents) represents the standard of care and is associated with an even worse prognosis in those patients who relapse with AML after transplantation.

The FLT3-TKI midostaurin has been approved for newly diagnosed AML patients with activating FLT3 mutations who receive intensive induction and subsequent consolidation chemotherapy including midostaurin maintenance restricted to patients who do not undergo allogeneic SCT. So far, there is no approval of FLT3-TKI treatment for patients with FLT3-mutated AML after allogeneic SCT. Recently, preliminary data of the RADIUS trial investigating midostaurin maintenance after allogeneic SCT could demonstrate the feasibility of midostaurin treatment in the setting of post-transplant AML patients. Importantly, only half of patients were able to complete 12 cycles of maintenance and in most cases midostaurin was prematurely ceased due to a higher rate of adverse events than expected. As a consequence of this clinical trial, there is a good rationale to investigate midostaurin maintenance after allogeneic SCT focusing on those AML patients with a high risk of hematologic relapse after transplantation.

In detail, MRD assessment provides a reliable method in the majority of patients with FLT3-mutated AML (e.g. by qPCR) to identify AML patients with the highest risk of relapse following allogeneic SCT. There are consistent data demonstrating that MRD positivity by means of NPM1 (Nuclophosphmin-1)mutation (i.e. 100 to 1000 copies of mutated NPM1 per 10,000 ABL (Abelson Murine Leukemia Viral Oncogene Homolog) transcripts or 1% to 10% NPM1/ABL, respectively, is associated with a 60-90% risk of hematologic relapse.

Thus, this clinically relevant subgroup of AML patients with activating FLT3 mutations who develop a molecular relapse or who are characterized by a persistent MRD positivity after intensive AML treatment represents the target population of this clinical trial. The rationale of this study is to treat AML patients with MRD positivity using single midostaurin treatment and to improve the clinical outcome of these patients by preventing hematologic relapse after allogeneic SCT by "targeted therapy" against activating FLT3 mutations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with molecular relapse or persistent molecular positivity of AML after allogeneic SCT (stem cell Transplantation)
* Detection of FLT3-ITD (Internal tandem duplication) or FLT3-TKD (tyrosine kinase domain) at primary diagnosis or at antecedent relapse of AML prior to allogeneic SCT
* Sensitive MRD assessment based on qPCR (e.g. by means of NPM1 mutations)
* absolute neutrophil count > 1,0 Gpt/L and Platelets > 50 Gpt/L
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* glomerular filtration rate > 30 ml/min and serum bilirubin < 1.5 x upper limit of normal
* Serum aspartate transaminase (AST) and/or alanine transaminase (ALT) ≤ 3.0 × ULN
* Normal serum levels of potassium, magnesium, and corrected calcium
* Written informed consent prior to any study procedures being performed
* Age ≥ 18 years

Exclusion Criteria:

* Acute promyelocytic leukemia (APL)
* Hematological relapse of AML
* Lack of a suitable MRD marker
* Impaired ejection fraction (LVEF) < 45%
* Patients with midostaurin treatment after allogeneic SCT or with ongoing TKI therapy < 4 weeks prior to inclusion
* Treatment with an investigational drug within 5 half-lives preceding the first dose of study medication
* History of acute or chronic pancreatitis
* Active and uncontrolled infections
* History of severe lung disease and/or relevant functional impairment
* Medical indication for treatment with strong CYP3A4 inhibitors (e.g. voriconazole, posaconazole, clarithromycin)
* Positive PCR for Human Immunodeficiency Virus (HIV) or Hepatitis B or C
* Patients unable to swallow medication
* Known hypersensitivity reaction to midostaurin or any excipient of midostaurin
* Concomitant medications with known induction of CYP3A4 isoenzyme unless they can be discontinued or replaced prior to enrollment
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who are pregnant or breast feeding, or females of reproductive potential not employing an effective method of birth control. Female patients must agree to an effective birth control throughout the study and for up to 4 months beyond.
* Other medical conditions (e.g. corrected QT interval prolongation) that might interfere with midostaurin treatment
* Substance abuse, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
proportion of patients without AML relapse | at 12 months after start of midostaurin treatment
  impact of midostaurin single treatment on Leukemia-free survival (LFS)

SECONDARY OUTCOMES:
number of patients with low MRD (Minimal Residual Disease) | at 3 months after start of midostaurin treatment
  molecular response to midostaurin treatment
Incidence of acute and chronic graft-versus-host disease (GvHD) | baseline and every 3 months until 12 months after start of midostaurin treatment
  Incidence of acute and chronic GvHD
Incidence of adverse events grade 3-5 of midostaurin after allogeneic SCT | baseline and every 3 months until 12 months after start of midostaurin treatment
  Incidence of adverse events grade 3-5
Next-generation sequencing analyses of FLT3-mutation | baseline and every 3 months until 12 months after start of midostaurin treatment
  mechanisms of primary or secondary resistance to midostaurin
quality of life assessment with certified "EORTC QLQ - C30 questionnaire" | baseline and every 3 months until 12 months after start of midostaurin treatment
  quality of life assessment with certified "EORTC QLQ - C30 questionnaire"

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Scholl, Prof. Dr., Principal Investigator — Jena University Hospital
Locations (4):
- Germany (4):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Leipzig AöR, Leipzig

IPD SHARING:
Plan to Share IPD: No